CLINICAL TRIAL: NCT03401814
Title: Imaging Response to Immunotherapy and Radiation Therapy in Patients With Liver Metastases
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sean S. Park, Radiation Oncology Consultant, Mayo Clinic
Other Study IDs: 17-009021; ROR1721 (Other: Mayo Clinic)
Record Dates: First submitted 2018-01-10; First posted 2018-01-17 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Liver Metastases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Magnetic Resonance Elastography — rapidly developing technology for quantitatively assessing the mechanical properties of tissue, using externally applied mechanical waves
  Other Names: MRE

SUMMARY:
Patients will be imaged with MRE at the time of the RT planning MRI, prior to the induction of RT and immunotherapy. Research imaging will be in addition to standard imaging studies performed at time points consistent with the standard of care (at the time of the RT planning MRI and the first clinical follow-up). An additional MRE exam will be performed at the end of treatment outside the standard of care imaging.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of solid cancers with the presence of one or more liver metastases
* Minimum metastasis diameter ≥ 2 cm
* Planning to receive radiation therapy with immunotherapy
* Willingness to participate in mandatory imaging studies at Mayo Clinic Rochester

Exclusion Criteria:

* Contraindications for MRI including claustrophobia, pace maker, metal implants, aneurism clips
* Patients who are not able to consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Radiation patients with liver metastases
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Quantify tissue mechanical properties of the liver and liver tumor using MRE in patients receiving radiation therapy + immunotherapy at baseline, mid-treatment and time of followup imaging determined by standard of care to assess response to therapy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sean Park, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials